CLINICAL TRIAL: NCT00586326
Title: MammoSite Radiation Therapy System (RTS) as the Sole Radiation Therapy Technique for Ductal Carcinoma In-Situ (DCIS)
Brief Title: MammoSite as Sole Radiation Therapy Technique for Ductal Carcinoma In-Situ
Acronym: DCIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-700
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: DCIS
Keywords: MammoSite; DCIS
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Women with DCIS (Experimental): Women with DCIS
  Interventions: Device: MammoSite Radiation Therapy System

INTERVENTIONS:
Device: MammoSite Radiation Therapy System — The MammoSite is a balloon catheter that is designed to position a radioactive source inside the lumpectomy cavity. The MammoSite applicator is inserted into the cavity created by the tumor removal surgery. The MammoSite applicator is then inflated and expands to fill the cavity.

SUMMARY:
This study has been designed to compile information on the efficacy of the MammoSite RTS providing sole radiation therapy for patients with pure DCIS.

DETAILED DESCRIPTION:
Data relevant to the evaluation of the efficacy and safety of the MammoSite RTS system in providing radiation therapy to patients with DCIS will be collected. The MammoSite is a radionuclide applicator designed to deliver internal radiation therapy (brachytherapy) in patients with breast tumors following breast tumor resection surgery (lumpectomy).

ELIGIBILITY:
Inclusion Criteria:

* Pre-Surgery:

  * Unicentric pure DCIS
  * Lesions should have a greatest dimension of 3 cm or less as determined by pre-surgery mammography and MRI
* Post-Surgery:

  * Negative histological margins confirmed prior to beginning radiation therapy.
  * Margins are positive if there is tumor at the inked margin.
  * Classified as low (NG1), intermediate (NG2) or high (NG3) nuclear grade DCIS, using the Philadelphia Consensus Conference Guidelines are eligible
  * Clinically node negative

Exclusion Criteria:

* Distance from the balloon surface to the surface of the skin < 5mm as determined by CT imaging.
* Distant metastases.
* Invasive or in-situ lobular carcinoma (post-surgery assessment).
* Nonepithelial breast malignancies such as sarcoma or lymphoma.
* DCIS that is multicentric in the ipsilateral breast.
* Pregnant or lactating.
* Prior non-hormonal therapy for the present breast cancer, including radiation therapy and/or chemotherapy.
* Collagen vascular diseases
* Coexisting medical conditions with life expectancy < 2 years.
* Serious psychiatric or addictive disorder
* Previously treated contralateral breast carcinoma
* Synchronous bilateral breast carcinoma.
* Other malignancy, except non-melanoma skin cancer, < 5 years prior to participation in the study; the disease free interval from any prior carcinoma must be continuous.
* Patients with diffuse disease

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2003-08; Primary Completion 2006-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Streeter, MD, Principal Investigator — University of Southern California
Locations (12):
- United States (12):
  - Arizona Oncology Services, Phoenix, Arizona
  - Daniel Freeman Hospital, Inglewood, California
  - University of Southern California, Los Angeles, California
  - Cedars Medical Center, Miami Beach, Florida
  - St. Agnes Hospital, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - NY Presbyterian, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - MD Anderson Cancer Clinic, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per the protocol, a total of 125 subjects were to be enrolled at 10-15 nationwide centers. A total of 133 subjects were enrolled at 12 nationwide centers. Patients with DCIS electing to undergo breast conserving therapy with radiation therapy were screened for enrollment.
Pre-assignment Details: Consented patients who were willing to enroll were evaluated prior to surgery. The lumpectomy was performed per the usual standard of care. The MammoSite applicator could be placed at the time of lumpectomy surgery or post-surgery in a separate procedure if adequate evacuated cavity was available as assessed by ultrasound.
Groups:
- Enrolled: Women with DCIS who were willing to enroll and consented
Period: Enrollment to Device Placement-Enrolled
Arm/Group | Enrolled
Started | 133
Completed | 118
Not Completed | 15
Not completed — Skin Distance | 6
Not completed — Cavity Conformance | 4
Not completed — Microinvasion | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1
Period: Device Placed toTreatment-ITT
Arm/Group | Enrolled
Started | 118
Completed | 100
Not Completed | 18
Not completed — Skin Distance | 7
Not completed — Cavity Conformance | 6
Not completed — Microinvasion | 1
Not completed — Positive Margins | 3
Not completed — Physician Decision | 1
Period: Treated Through 5-yr Follow Up-Treated
Arm/Group | Enrolled
Started | 100
Completed | 74
Not Completed | 26
Not completed — Clinical Reason | 1
Not completed — Death | 2
Not completed — Medical Reason | 2
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 14
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- Treated: Subjects enrolled with device placed and treated with partial breast irradiation
Arm/Group | Treated
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 69
  >=65 years | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Local Control Rate for Follow-up Period of 5 Years.
Description: Failure of local control was defined as a histologically confirmed recurrence (invasive or non-invasive) within the prescription isodose volume. All recurrences were to have histological evaluation per the protocol; however, the case report forms did not provide space for this data to be captured. Ipsilateral axillary, infraclavicular, internal mammary, or supraclavicular recurrence or distant metastases were not considered treatment failures unless accompanied by ipsilateral breast failure.
Time Frame: Data collected at the time of implant, radiation therapy, and at the patient's 3 month, 6 month, 1 year, 2 year, 3 year, 4 year and 5 year follow-up visits.
Measure: Number; unit: percentage of subjects
Arm/Group | Treated
Number analyzed (Participants) | 100
percentage of subjects | 99

2. Secondary Outcome: Overall Survival
Time Frame: At 5 Years
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Treated
Number analyzed (Participants) | 100
participants | 97.7 [94.6 to 100.0]

3. Secondary Outcome: Cause Specific Survival
Time Frame: At 5 Years
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Treated
Number analyzed (Participants) | 100
participants | 100.0 [100.0 to 100.0]

4. Secondary Outcome: Disease Free Survival
Time Frame: At 5 Years
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Treated
Number analyzed (Participants) | 100
participants | 98.9 [96.7 to 100.0]

5. Secondary Outcome: Cosmetic Evaluations Over Time
Description: As assessed using the four category Harvard Scale for subjects with an evaluation at the 5 year timepoint
Time Frame: At 5 Years
Population: Subjects with Cosmetic Evaluation at 5 Years
Measure: Number; unit: percentage of subjects
Groups:
- Excellent: Subjects enrolled with device placed and treated with partial breast irradiation who had the cosmetic evaluation scored as 'Excellent' at 5 years
- Good: Subjects enrolled with device placed and treated with partial breast irradiation who had the cosmetic evaluation scored as 'Good' at 5 years
- Fair: Subjects enrolled with device placed and treated with partial breast irradiation who had the cosmetic evaluation scored as 'Fair' at 5 years
- Poor: Subjects enrolled with device placed and treated with partial breast irradiation who had the cosmetic evaluation scored as 'Poor' at 5 years
Arm/Group | Excellent | Good | Fair | Poor
Number analyzed (Participants) | 47 | 47 | 47 | 47
percentage of subjects | 42.6 | 44.7 | 12.8 | 0.0

ADVERSE EVENTS:
Groups:
- Intent to Treat: Enrolled subjects with MammoSite device placed
Arm/Group | Intent to Treat
Serious Adverse Events (participants affected / at risk) | 6/118
Other Adverse Events (participants affected / at risk) | 97/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent to Treat (N=118)
Cerebral Vascular Accident (Vascular disorders) | 2 (2) — Subject 09-001 suffered a cerebral vascular accident (CVA) and Subject 09-014 experienced a CVA. Both were determined to be 'Not Related'.
Lung cancer with metastases to the brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Subject 09-013 developed lung cancer with metastases to the brain and subsequently died. The event was determined to be 'Not Related'.
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) — Subject 01-002 had abnormal uterine bleeding requiring hysterectomy. The event was determined to be 'Not Related'.
Cellulitis (Infections and infestations) | 1 (1) — Subject 11-011 was admitted to the hospital for evaluation of pain, swelling, fever & chills and was diagnosed with cellulitis & started on IV antibiotics. Event was believed unlikely related & was reported as serious due to hospitalization.
Infection (Infections and infestations) | 1 (1) — One subject in the ITT population experienced an event of infection (Subject 11-014). This event was reported as serious, probably related to the device and after treatment, resolved without sequelae.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intent to Treat (N=118)
Seroma (Injury, poisoning and procedural complications) | 38
Infection (Infections and infestations) | 4
Fat Necrosis (General disorders) | 14
Telangiectasia (Skin and subcutaneous tissue disorders) | 22
Fibrosis (General disorders) | 41
Induration (General disorders) | 30
Breast Pain (Reproductive system and breast disorders) | 29
Retraction (Skin and subcutaneous tissue disorders) | 9
Radiation Dermatitis (Injury, poisoning and procedural complications) | 7
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 19
Rib pain (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days